CLINICAL TRIAL: NCT03930719
Title: Evaluation of Delirium Screening Tools for the Detection of Post-stroke Delirium
Brief Title: Post-stroke Delirium Screening
Acronym: PSD Screen
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 031-19
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Delirium; Ischemic Stroke; Transient Ischemic Attack
Keywords: stroke; delirium; screening tool
MeSH Terms: conditions — Delirium; Ischemic Stroke; Ischemic Attack, Transient; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSD: Patients fulfilling DSM-5 criteria of PSD within 7 days of admission.
  Interventions: Diagnostic Test: Stroke screening tools
- No PSD: Patients NOT fulfilling DSM-5 criteria of PSD within 7 days of admission.
  Interventions: Diagnostic Test: Stroke screening tools

INTERVENTIONS:
Diagnostic Test: Stroke screening tools — Patients are evaluated for the presence of PSD using DSM-5 criteria ("gold standard"). Established delirium detection tools are evaluated for their diagnostic accuracy compared to the gold standard.

SUMMARY:
For a long time, delirium was considered a merely temporary dysfunction of the brain. Today, it is established that it is a brain disease associated with network dysfunction, neuroinflammation and impaired transmitter homeostasis in a multicausal model. Following an episode of delirium, many patients do not return to their prior level of cognitive and functional performance. In particular, failed or delayed diagnosis with consecutive inadequate therapy contribute to the development of long-term cognitive decline that may ultimately lead to long-term care. Stroke patients are a particularly common delirium-affected population (10-46% depending on severity). Despite the frequency and clinical relevance of delirium in stroke patients, diagnostic characteristics of common screening methods are unknown. Similarly, the clinical phenotype and risk factors of patients who develop delirium have not been adequately described.

This study primarily aims to evaluate the diagnostic properties of established screening tools for delirium in a prospective cohort of well-characterised patients following ischemic cerebral events (either transient or manifest stroke). Secondary outcome criteria include predictors of post-stroke delirium (PSD) such as stroke location and size, pre-stroke cognitive functioning, ability to participate in daily routine activities and medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* stroke unit admission for a high-risk transient ischemic attack (ABCD2 score >= 6) or stroke within the last 24 hours

Exclusion Criteria:

* hemorrhagic stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient admitted to the emergency department for a suspected ischemic cerebrovascular event is eligible to participate. A neurologist must then confirm the diagnosis and necessity for stroke unit monitoring.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of established delirium detection tools as compared to Diagnostic and Statistical Manual - 5th Version (DSM-5) criteria | two times daily for 7 days
  Binary outcomes of delirium screening tests will be compared, i.e. if they characterize an individual patient as delirious at any of two time points during the 7 day observation period. Instruments include: Nursing Delirium Screening Scale (Nu-DESC), Confusion Assessment Method (CAM), rapid assessment test for delirium (4-AT). Binary outcomes ("yes" or "no" according to each of the scales) are then aggregated in one test that compares the observed frequency of delirious patients (according the above mentioned tests) with the actual number of delirious patients as assessed by the DSM-5 standard.

SECONDARY OUTCOMES:
PSD prevalence | three times daily for 7 days
  DSM-5 criteria and chart review are used to assess the occurence of PSD among included patients over the complete study period
pre-stroke modified Rankin Scale | once on admission
  functional status before stroke
pre-stroke Barthel Index | once on admission
  ability to take care of personal daily routine before stroke
pre-stroke Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | once on admission
  cognitive impairment before stroke
pre-stroke Groningen Frailty Index (GFI) | once on admission
  presence of a frailty syndrome before stroke
National Institutes of Health Stroke Scale (NIHSS) | three times daily for three days starting on the day of admission
  estimate of clinical stroke severity
Critical Care Pain Observation Tool (CPOT) | once daily for three days starting on the day of admission
  pain during stroke unit treatment
Stroke location - clinical (classification of the OxfordshireCommunity Stroke Project (OCSP)) | once on admission
  clinical characterisation based on phenotype as either total anterior, partial anterior, partial posterior or lacunar stroke
Stroke location - imaging (based on an atlas of anatomical regions of the human brain (aal MNI V4)) | once on admission
  in patients with imaging of the definite stroke location, differences of mean locations between groups will be calculated

OTHER OUTCOMES:
demographic data | once on admission
  exploratory outcome required to adjust for confounding variates such as age, socioeconomic status and education
complications during stroke unit treatment | continuously during the study period and up to 7 days
  any complication that arises during the study period (e.g. pneumonia, dysphagia)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fleischmann, MD, Principal Investigator — Department of Neurology
Locations (1):
- Department of Neurology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleischmann R, Warwas S, Andrasch T, Kunz R, Witt C, Mengel A, von Sarnowski B. Course and Recognition of Poststroke Delirium: A Prospective Noninferiority Trial of Delirium Screening Tools. Stroke. 2021 Jan;52(2):471-478. doi: 10.1161/STROKEAHA.120.031019. Epub 2020 Dec 31. PMID 33380165